CLINICAL TRIAL: NCT06655142
Title: Prospective Matched Control Feasibility Study to Determine the Capacity of the Onco-Seraph 100 Microbind® Affinity Blood Filter ( ONCObind Procedure) to Remove Circulating Tumor Cells From the Blood in Patients With Either Metastatic Pancreatic Adenocarcinoma or Metastatic Colorectal Carcinoma
Brief Title: OSCAR II STUDY - The ONCObind CTC Removal Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ExThera Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Onco-Seraph-US23-002
Record Dates: First submitted 2024-10-19; First posted 2024-10-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma (mPDAC); Metastatic Colorectal Carcinoma (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Study patients will be assigned to receive procedure with the investigational device (ONCObind) and will be matched with site specific controls. 60 with ONCObind procedure and 60 Controlled
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ONCObind (Onco-Seraph) 100 Filter is a single use (Experimental): The ONCObind Filter is a single use, disposable column packed with ultra-high molecular weight polyethylene beads which have been modified to contain endpoint attached heparin on the surface. The devices are sterilized using a standard ethylene oxide cycle, following ISO 11135-1:2007. Chemical Indicator labels are located near the product label. ONCObind is part of the Seraph platform technology that was also developed as an extracorporeal broad-spectrum sorbent hemoperfusion device for reduction of pathogens from the bloodstream.
  Interventions: Device: ONCObind (Onco-Seraph) 100 Filter
- Matched Controls (Other): Study patients will be assigned to receive procedure with the investigational device (ONCObind) and will be matched with 60 site specific controls, 30 PDAC and 30 CRC.
  Interventions: Other: Matched Controls

INTERVENTIONS:
Device: ONCObind (Onco-Seraph) 100 Filter — The ONCObind Microbind® Affinity Blood Filter ( ONCObind) manufactured by ExThera Medical Corporation in Martinez, CA. The ONCObind filter has been designed and manufactured to reduce residual risks as much as possible to ensure safe usage. Literature search results concluded that heparin-coated medical devices are safe and decrease platelet adhesion without affecting the adsorption of major adhesive proteins. Literature search yielded over 60 publications and 500 treated patients with Seraph platform technology for pathogen removals without and significant safety concern. The achieved results from the above-mentioned testing and studies support the performance and safety of ONCObind consistent with the intended use. ExThera Medical concludes that the known and potential benefits of ONCObind, when used to treat patients with PDAC, outweigh the known and potential risks when used according to the intended use.
  Arms: ONCObind (Onco-Seraph) 100 Filter is a single use
Other: Matched Controls — Study patients will be assigned to receive procedure with the investigational device (ONCObind) and will be matched with 60 site specific controls, 30 PDAC and 30 CRC.
  Arms: Matched Controls

SUMMARY:
This study is a Prospective Single Arm, dual cohort Open Label Feasibility trial to evaluate the initial safety and signal of efficacy of a novel extracorporeal blood purification (EBP) procedure in either mPDAC or mCRC refractory to systemic therapy. Site selection will be dependent upon the site's familiarity with extracorporeal blood purification platforms as well as the diagnosis and management of mPDAC and mCRC. Adults (18 years old and older, ECOG PS of equal or less than 2) with a diagnosis of either mPDAC as defined histologically (microscopically) as a "pancreatobiliary type" adenocarcinoma who experienced disease progression or not tolerating fluoropyrimidine-, oxaliplatin- and irinotecan- based regimens or prior treatment with gemcitabine and nab-paclitaxel or are not candidates for chemotherapy or mCRC patients who experienced disease progression on 5-fluorouracil (5-FU), capecitabine, oxaliplatin and irinotecan as FOLFIRI and/or FOLFOX and/or XELOX and/or XELIR and/or FOLFOXIRI/FOLFIRINOX or who are not candidates for chemotherapy with at least 5 cells/mL CTCs in peripheral blood and/or portal vein.

DETAILED DESCRIPTION:
Study Intervention: All study patients will be assigned to receive procedure with the investigational device (ONCObind ) Study Duration: Our target enrollment is 30 patients with mPDAC and 30 patients with mCRC. The study will last for up to two years. Interim analyses will determine early stopping for safety. This is detailed in Section 22: Data Safety Monitoring Board (DSMB). Furthermore, as the safety and effectiveness of the experimental use of the ONCObind device for treatment of patients with mPDAC and/or mCRC is unknown, patients will be followed for up to 5 years to inform oncological outcomes.

Procedure Setting: Extracorporeal blood purification utilizing ONCObind can be performed either on an outpatient or an in-patient basis as HD/CRRT procedure is performed routinely in both settings. Whether the procedure will be performed in a setting of an outpatient or in-patient setting would mainly depend on the personalized approach that the Site Investigator choses related to individual patient enrolled in the study. Location of the ONCObind treatment will be recorded, and data analysis will include consideration of the setting as it relates to study endpoints. If the Study Procedure is implemented in an outpatient setting, the subject will be monitored for up to 4 hours post procedure per PI discretion.

Procedure Duration for ONCObind : A sufficient blood flow rate and exposure of patient's blood to the ONCObind adsorption media was initially established based on the experience in implementing procedure in patients with blood stream infections. However, target procedure duration is further optimized based on data collected in EU oncology patients as listed below:

the average procedure duration and blood flow rates targeted in patients with blood stream infections or oncology are as follows:

* At an average blood flow of 350mL/min, this would translate to approximately 5 hours of procedure time for patients with blood stream infection or 2.0 hours for an oncology patient; an average of 200mL/min translates to a procedure time of 8 hours for blood stream infection or 3.5 hrs for oncology patient.
* OSCAR I 1st Stage: Study Procedure will occur only once, followed by weekly follow up visits through day 28, followed by monthly follow up through Day 60
* OSCAR II 2nd Stage: Study Procedure s will occur up to 3-5 times for the first week followed by 1-3treatments through week 4, for a total of up to 8 treatments over the first 28 days of study participation. Study treatments will continue every 4 weeks (+/- 1 week) from week 5 through week 26.
* Study Procedure(s) will be held, if subjects are hemodynamically unstable and unable to tolerate extracorporeal procedure (defined as MAP<65 and or sustained hypotension at enrollment as defined by two readings with systolic blood pressure (SBP) measurements below 100 mmHg or diastolic blood pressure (DBP) measurements below 50 mmHg. The measurements must be performed thirty minutes from one another, and the Subject must be resting for at least 5 minutes prior to obtaining each measurement. (If the first reading includes a SBP greater than 100 mmHg and a DBP greater than 50 mmHg, the second reading does not need to be taken).

Subjects will be assessed per study visits and as part of routine, standard of care for mPDAC or mCRC. All subjects enrolled in this study will undergo clinical efficacy, safety, and laboratory assessments. Blood, and clinical data collection samples will be obtained at Screening, Induction Phase, and Procedure Follow up Phase in accordance to Schedule of Events. . Demographic and baseline clinical parameters will be recorded at the time of enrollment. Pertinent clinical parameters will be recorded in accordance to Schedule of Events . Outcomes data will be recorded on in accordance to Schedule of Events . Subject status will be in accordance to Schedule of Events to include adverse event evaluation and a targeted medication review. Survival follow-up will be assessed at 60, 120, 180 and 210 days after enrollment and/or at the time of death.

Patients will receive standard of care follow-up for up to 5 years and this data collected will be made available for FDA review.

A subset of the protocol team will review Grade 3 and 4 adverse event or serious adverse event (AE / SAE) data every 2 weeks. If there is a pattern of unexpected AEs that is out of proportion to the current understanding of the natural history of the disease, the DSMB will be asked to review un-blinded safety data in an ad hoc meeting. If an ad hoc meeting of the DSMB is convened to review a serious, device-related adverse event, enrollment will be halted pending the DSMB review to ensure subject safety in the trial. The DSMB will review the event to ensure subject safety. After the review, the DSMB will determine if enrollment may resume.

The DSMB will conduct an interim analysis after the enrollment of 10 subjects in each mPDAC and mCRC cohort to evaluate for safety and efficacy prior to completion of enrollment (n=30 for each cohort) (as detailed in Data Safety Monitoring Board (DSMB) and will be available for ad hoc reviews for safety concerns as described above. As stated above, enrollment will be halted pending the convening of an ad hoc DSMB meeting to review a serious, device-related adverse event. The DSMB will review the event to ensure subject safety in the trial. The DSMB will determine if enrollment may resume. The DSMB may recommend temporary or permanent cessation of enrollment based on their safety reviews.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet all of the following criteria:

1. Patients ≥ 18 years of age with

   1. mPDAC cohort: Metastatic pancreatic ductal cancer who experienced disease progression or not tolerating fluoropyrimidine-, oxaliplatin- and irinotecan- based regimens or prior treatment with gemcitabine and nab-paclitaxel or are not a candidate for chemotherapy
   2. mCRC Cohort : Metastatic CRC who experienced disease progression on 5-fluorouracil (5-FU), capecitabine, oxaliplatin and irinotecan as FOLFIRI and/or FOLFOX and/or XELOX and/or XELIRI and/or FOLFOXIRI/FOLFIRINOX or who are not candidates for chemotherapy.
2. Patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) scores of 2 or less.
3. Patient or legally authorized representative is willing and able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
4. Patients with a CTC concentration of at least 5 cells/mL
5. Must be willing to provide blood samples for prospective tumor molecular profiling and exploratory analyses.
6. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
7. Patients must be of non-childbearing potential or using a medically acceptable contraceptive regimen. Effective contraception includes surgical sterilization (e.g., vasectomy, tubal ligation), two forms of barrier methods (e.g., condom, diaphragm) used with spermicide, IUDs.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnant or breast feeding
2. Patients who cannot tolerate the placement of a tunneled catheter for vascular access to enable extracorporeal treatment.
3. Patients with a history of heparin induced thrombocytopenia (HIT).
4. Patients with known allergy to heparin sodium.
5. High risk of bleeding (platelet count <50mm3 or International Normalized Ratio (INR) >1.5)
6. Hemodynamic instability and inability to tolerate extracorporeal therapy (defined as MAP<65 despite fluids and vasopressors and or sustained hypotension at enrollment as defined by two readings with systolic blood pressure (SBP) measurements below 100 mmHg or diastolic blood pressure (DBP) measurements below 50 mmHg. The measurements must be performed thirty minutes from one another, and the Subject must be resting for at least 5 minutes prior to obtaining each measurement. (If the first reading includes a SBP greater than 100 mmHg and a DBP greater than 50 mmHg, the second reading does not need to be taken).
7. Uncontrolled hypertension despite optimal management (systolic blood pressure >180mmHg
8. Ongoing uncontrolled, serious infection.
9. Renal failure requiring dialysis.
10. Patients with a life expectancy of less than 30 days.
11. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to initiation of treatment on this study.
12. Concurrent participation in any interventional clinical trial or has been previously entered in this trial.
13. The Patient is a prisoner or member of a different vulnerable population that should not be included in the study per the investigator.
14. Unable to obtain informed consent from either patient or legally authorized representative (LAR)
15. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedure-emergent adverse events (AEs) graded using the NCI CTCAE Version 5.0 | 210 days
  Incidence of procedure-emergent adverse events (AEs) graded using the NCI CTCAE Version 5.0
Incidence of procedure-emergent serious adverse events (SAEs) graded using the NCI CTCAE Version 5.0 | 210 days
  Incidence of procedure-emergent serious adverse events (SAEs) graded using the NCI CTCAE Version 5.0
Evaluation of Survival | 60, 120, 180 and 210 days
  Survival follow-up will be assessed after enrollment (vital status check)
Change in CTC Concentration | 180 days
  The change in CTC concentration from baseline to the end of the induction series as well as 180 days after baseline of Extracorporeal Procedure (ECPs) with ONCObind
Capacity for the ONCObind filter to remove circulating tumor cells | 60 days
  Capacity for the ONCObind filter to remove circulating tumor cells (CTCs) when compared to baseline
Evaluate the Quality of Life (QOL) | 210 days
  To evaluate the Quality of Life from baseline to end of study using the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Lakhmir Chawla, M.D., Principal Investigator — ExThera Medical

IPD SHARING:
Plan to Share IPD: No
Following completion of the study, results of this research will be in a scientific journal. Data will be available immediately following publication, with no end date, with data sharing at the discretion of the Sponsor.